CLINICAL TRIAL: NCT03011372
Title: A Phase 2, Open-Label, Monotherapy, Multicenter Study to Evaluate the Efficacy and Safety of Pemigatinib (INCB054828) in Subjects With Myeloid/Lymphoid Neoplasms With FGFR1 Rearrangement - (FIGHT-203)
Brief Title: A Study to Evaluate the Efficacy and Safety of Pemigatinib (INCB054828) in Subjects With Myeloid/Lymphoid Neoplasms With FGFR1 Rearrangement - (FIGHT-203)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 54828-203; 2016-002596-10 (EudraCT Number)
Expanded Access: NCT03906357 (No longer available)
Record Dates: First submitted 2017-01-04; First posted 2017-01-05 (Estimated); Results first posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: MPN (Myeloproliferative Neoplasms)
Keywords: Myeloid neoplasm; fibroblast growth factor receptor inhibitor; FGFR1 rearrangement; 8p11; eosinophilia; eosinophilic syndrome; Lymphoid neoplasm
MeSH Terms: conditions — Myeloproliferative Disorders; Eosinophilia | interventions — pemigatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pemigatinib (Experimental)
  Interventions: Drug: Pemigatinib

INTERVENTIONS:
Drug: Pemigatinib — Pemigatinib once a day by mouth for 2 consecutive weeks and 1 week off therapy.
  Participants will receive either the intermittent dose (as written) or continuous dosing.
  Other Names: INCB054828

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of pemigatinib (INCB054828) in subjects with myeloid/lymphoid neoplasms with fibroblast growth factor receptor (FGFR) 1 rearrangement.

ELIGIBILITY:
Inclusion Criteria:

* Documented lymphoid or myeloid neoplasm with 8p11 rearrangement known to lead to FGFR1 activation, based on standard diagnostic cytogenetic evaluation performed locally, before signing informed consent for this study.
* Eligible subjects must:

  * Have relapsed after stem cell transplantation or after other disease modifying therapy, OR
  * Not be current candidates for stem cell transplantation or other disease modifying therapies.
* Note: All relapsed/refractory subjects must have evidence of either cytogenetic or hematological disease and have no evidence of residual toxicity (eg, graft-versus-host disease requiring treatment).
* Life expectancy ≥ 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.

Exclusion Criteria:

* Prior receipt of a selective FGFR inhibitor.
* History and/or current evidence of ectopic mineralization/calcification, including but not limited to soft tissue, kidneys, intestine, myocardia, or lung, except calcified lymph nodes and asymptomatic arterial or cartilage/tendon calcifications.
* Current evidence of corneal disorder/keratopathy, including but not limited to bullous/band keratopathy, corneal abrasion, inflammation/ulceration, and keratoconjunctivitis, as confirmed by ophthalmologic examination.
* Use of any potent cytochrome P450 3A4 inhibitors or inducers within 14 days or 5 half-lives (whichever is shorter) before the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philomena Collucci, MD, Study Director — Incyte Corporation
Locations (33):
- United States (9):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - City of Hope National Medical Center, Duarte, California
  - Stanford Cancer Institute, Stanford, California
  - Emory University - Winship Cancer Institute, Atlanta, Georgia
  - Franciscan St. Francis Health, Indianapolis, Indiana
  - Washington University School of Medicine, St Louis, Missouri
  - Weill Cornell Medical Centers, New York, New York
  - Md Anderson Cancer Center, Houston, Texas
  - University of Utah, Salt Lake City, Utah
- Austria (3):
  - Ordensklinikum Krankenhaus Der Barmherzigen Schwestern Linz, Linz
  - Medical University of Vienna, Vienna
  - Iii Med. Abteilung For Hematologie and Onkologie Hanuscfhkrankenhaus, Vienna
- Universitair Ziekenhuis (Uz) Leuven, Leuven, Belgium
- Princess Margaret Cancer Center, Toronto, Ontario, Canada
- France (4):
  - Centre Leon Berard, Lyon
  - Chu de Nice - Hospital L Archet, Nice
  - Hospital Saint Louis, Paris
  - Universitaire Du Cancer de Toulouse Institut Claudius Regaud Iuct-Oncopole, Toulouse
- Germany (6):
  - University Medical Center Rwth Aachen, Aachen
  - Universitatsklinikum Halle (Saale), Halle
  - Universitatsklinikum Jena, Jena
  - Universitatsklinikum Leipzig, Leipzig
  - University Hospital Mannheim, Mannheim
  - Johannes Wesling Klinikum Minden, Minden
- Italy (2):
  - Ospedale Papa Giovanni Xxiii, Bergamo
  - Azienda Ospedaliero-Universitaria Careggi (Aouc), Florence
- Japan (2):
  - Kindai University Hospital, Osaka
  - Ntt Medical Center Tokyo, Tokyo
- Hospital Clinico Universitario de Valencia, Valencia, Spain
- Switzerland (2):
  - Inselspital - Universitaetsspital Bern, Bern
  - Universitatsspital Zurich, Zurich
- United Kingdom (2):
  - Guys and St Thomas Nhs Foundation Trust, London
  - Oxford University Hospitals Nhs Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- [Derived] Al-Bazaz M, Forstreuter A, Hammada I, Hille J, Wagner JN, Reinert J, Wehrhahn J, Bokemeyer C, Fiedler W. Acute Lymphoblastic Leukemia Characterized by Rare BCR::FGFR1 Translocation: A Case Report With Literature Review. Case Rep Hematol. 2025 Oct 23;2025:8892036. doi: 10.1155/crh/8892036. eCollection 2025. PMID 41180818
- [Derived] Verstovsek S, Kiladjian JJ, Vannucchi AM, Patel JL, Rambaldi A, Shomali WE, Oh ST, Usuki K, Harrison CN, Ritchie EK, Akard LP, Hernandez-Boluda JC, Huguet F, Colucci P, Zhen H, Oliveira N, Gilmartin A, Langford C, George TI, Reiter A, Gotlib J. Pemigatinib for Myeloid/Lymphoid Neoplasms with FGFR1 Rearrangement. NEJM Evid. 2025 Sep;4(9):EVIDoa2500017. doi: 10.1056/EVIDoa2500017. Epub 2025 Aug 26. PMID 40856555
- [Derived] Subbiah V, Burris HA 3rd, Kurzrock R. Revolutionizing cancer drug development: Harnessing the potential of basket trials. Cancer. 2024 Jan;130(2):186-200. doi: 10.1002/cncr.35085. Epub 2023 Nov 7. PMID 37934000

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted at 21 study centers in Belgium, Canada, France, Germany, Italy, Japan, Spain, United Kingdom, and the United States.
Groups:
- Pemigatinib 13.5 mg: Pemigatinib 13.5 milligrams (mg) was self-administered once daily (QD) as oral tablets on an intermittent dosing (ID) schedule or continuous dosing (CD) schedule. Participants started pemigatinib 13.5 mg on the ID schedule (i.e., 2 weeks on/1 week off) as per the initial Protocol and on the CD schedule in 21-day cycles following a Protocol amendment.
Period: Overall Study
Arm/Group | Pemigatinib 13.5 mg
Started | 47
Completed | 0
Not Completed | 47
Not completed — Death | 16
Not completed — Lost to Follow-up | 2
Not completed — Sponsor Decision | 17
Not completed — Withdrawal by Subject | 7
Not completed — Moved to Commercial Supply of Investigational Drug | 2
Not completed — Received First Dose of Chemotherapy for Stem Cell Transplant | 1
Not completed — Sponsor's Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Pemigatinib 13.5 mg
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (13.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 30
  Black or African American | 4
  Asian | 4
  Missing | 5
  Not Provided | 2
  White/Caucasian and American-Indian Alaska Native | 1
  African | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 33
  Not Reported | 8
  Unknown | 1
  Captured as "Other" in Database | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Complete Response (CR) as Determined by Investigator Assessment According to the Response Criteria for Myeloid/Lymphoid Neoplasms With FGFR1 Rearrangement
Description: CR was defined as the presence of all of the following improvements: (1) bone marrow: ≤5% myeloblasts (including monocytic blast equivalent) and no lymphoblasts, with normal maturation of all cell lines, and return to age-adjusted normal cellularity; (2) osteomyelofibrosis absent or equal to "mild reticulin fibrosis" (Grade 1 or less fibrosis); (3) peripheral blood: white blood cells (WBC) ≤10 x 10^9 cells/Liter (L); hemoglobin (Hgb) ≥11 grams per deciliter (g/dL); platelets ≥100 x 10^9/L and ≤450 x 10^9/L; neutrophils ≥1.0 x 10^9/L; blasts = 0%; neutrophil precursors reduced to ≤2%; monocytes ≤1 x 10^9/L; eosinophils ≤0.5 x 10^9/L; (4) extramedullary disease: complete resolution of extramedullary disease present before therapy (e.g., lymphadenopathy), including palpable hepatosplenomegaly. Persistent low-level dysplasia was permitted given subjectivity of assignment of dysplasia. Response criteria by investigator assessment were the same for chronic phase (CP) and blast phase (BP).
Time Frame: up to 2513 days (120 21-day treatment cycles)
Population: Full Efficacy-Evaluable Population: all enrolled participants with an FGFR1 rearrangement and who received at least 1 dose of study drug. For this report, the full EEP included both previously treated and treatment-naive participants. Confidence intervals were calculated based on the exact method for binomial distribution.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemigatinib 13.5 mg
Number analyzed (Participants) | 45
percentage of participants | 68.9 [53.35 to 81.83]

2. Other Pre Specified Outcome: Percentage of Participants Who Achieved CR as Determined by Central Review Committee (CRC) Assessment
Description: In addition, responses were assessed by CRC based on Myeloid/Lymphoid Neoplasm International Working Group (MLN IWG) response criteria for myeloid/lymphoid neoplasms with eosinophilia and tyrosine kinase gene fusions.
Time Frame: up to 2513 days (120 21-day treatment cycles)
Population: Full Efficacy-Evaluable Population. Confidence intervals were calculated based on the exact method for binomial distribution.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemigatinib 13.5 mg
Number analyzed (Participants) | 45
percentage of participants | 68.9 [53.35 to 81.83]

3. Secondary Outcome: Percentage of Participants Who Achieved a Best Overall Response of Complete Response (CR) or Partial Response (PR) as Determined by Investigator Assessment According to the Response Criteria for Myeloid/Lymphoid Neoplasms With FGFR1 Rearrangement
Description: CR=all of the following improvements: (1) bone marrow: ≤5% myeloblasts (including monocytic blast equivalent) and no lymphoblasts, with normal maturation of all cell lines, and return to age-adjusted normal cellularity; (2) osteomyelofibrosis absent/equal to "mild reticulin fibrosis"; (3) WBC ≤10 x 10^9 cells/L; Hgb ≥11 g/dL; platelets ≥100 x 10^9/L, ≤450 x 10^9/L; neutrophils ≥1.0 x 10^9/L; blasts=0%; neutrophil precursors reduced to ≤2%; monocytes ≤1 x 10^9/L; eosinophils ≤0.5 x 10^9/L; (4) extramedullary disease: complete resolution of extramedullary disease present pre-therapy, including palpable hepatosplenomegaly. Persistent low-level dysplasia was permitted. PR=all of the following improvements: (1) reduction of bone marrow blasts/blast equivalents by 50%, but remaining >5% of cellularity (except in cases with ≤5% bone marrow blasts at baseline); (2) normalization of peripheral blood indices per CR Criterion 3; (3) extra medullary disease response of CMR/CR or PMR/PR.
Time Frame: up to 2513 days (120 21-day treatment cycles)
Population: Full Efficacy-Evaluable Population. Confidence intervals were calculated based on the exact method for binomial distribution. CMR=complete metabolic response; PMR=partial metabolic response. Response criteria by investigator assessment were the same for chronic phase (CP) and blast phase (BP).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemigatinib 13.5 mg
Number analyzed (Participants) | 45
percentage of participants | 77.8 [62.91 to 88.80]

4. Other Pre Specified Outcome: Percentage of Participants Who Achieved a Best Overall Response of CR or PR as Determined by CRC Assessment
Description: In addition, responses were assessed by CRC based on MLN IWG response criteria for myeloid/lymphoid neoplasms with eosinophilia and tyrosine kinase gene fusions.
Time Frame: up to 2513 days (120 21-day treatment cycles)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemigatinib 13.5 mg
Number analyzed (Participants) | 45
percentage of participants | 75.6 [60.46 to 87.12]

5. Secondary Outcome: Percentage of Participants Who Achieved a Complete Cytogenetic Response (CCyR) as Assessed by Local Analysis and Investigator Evaluation
Description: CCyR was defined as 0% 8p11 translocated metaphases as seen on classic karyotyping with minimal of 20 metaphases, or fluorescence in situ hybridization (FISH). Loss of cytogenetic burden of disease (via FISH or classic karyotyping) was required to reach CCyR.
Time Frame: up to 2513 days (120 21-day treatment cycles)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemigatinib 13.5 mg
Number analyzed (Participants) | 45
percentage of participants | 73.3 [58.06 to 85.40]

6. Other Pre Specified Outcome: Percentage of Participants Who Achieved a CCyR as Assessed by CRC Assessment
Description: as for outcome 4
Time Frame: up to 2513 days (120 21-day treatment cycles)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemigatinib 13.5 mg
Number analyzed (Participants) | 45
percentage of participants | 73.3 [58.06 to 85.40]

7. Secondary Outcome: Percentage of Participants Who Achieved a Partial Cytogenetic Response (PCyR) as Assessed by Local Analysis and Investigator Evaluation
Description: PCyR was defined as the decrease from baseline of 50% or more 8p11 translocated metaphases as seen on classic karyotyping with minimal of 20 metaphases, or FISH.
Time Frame: up to 2513 days (120 21-day treatment cycles)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemigatinib 13.5 mg
Number analyzed (Participants) | 45
percentage of participants | 8.9 [2.48 to 21.22]

8. Secondary Outcome: Percentage of Participants Who Achieved a PCyR as Assessed by CRC Assessment
Description: as for outcome 4
Time Frame: up to 2513 days (120 21-day treatment cycles)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemigatinib 13.5 mg
Number analyzed (Participants) | 45
percentage of participants | 15.6 [6.49 to 29.46]

9. Secondary Outcome: Duration of Complete Response
Description: Duration of complete response was defined as the time from the first assessment of complete response to the earlier of the date of first worsening assessment after complete response or death due to any cause
Time Frame: up to 2513 days (120 21-day treatment cycles)
Population: Full Efficacy-Evaluable Population. Only participants with a complete response were analyzed. Confidence intervals were calculated using the Brookmeyer and Crowley's method.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemigatinib 13.5 mg
Number analyzed (Participants) | 31
months
  Investigator assessment | 53.29 [12.22 to NA] — The upper limit of the confidence interval was not estimable because too few participants had worsening assessment after response or death.
  CRC assessment | NA [27.86 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants had worsening assessment after response or death.

10. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time from the first assessment of complete response or partial response to the earlier of the date of first worsening assessment after response or death due to any cause.
Time Frame: up to 2513 days (120 21-day treatment cycles)
Population: Full Efficacy-Evaluable Population. Only participants with complete response or partial response were analyzed. Confidence intervals were calculated based on the exact method for binomial distribution.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemigatinib 13.5 mg
Number analyzed (Participants) | 45
months
  Investigator assessment: number analyzed (Participants) | 35
  Investigator assessment | 53.29 [15.51 to NA] — The upper limit of the confidence interval was not estimable because too few participants had events of loss of response (disease progression) or death.
  CRC assessment: number analyzed (Participants) | 34
  CRC assessment | NA [27.86 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants had events of loss of response (disease progression) or death.

11. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from the first date of taking study drug until the date of disease progression or until death due to any cause, whichever was earlier. Disease progression was defined as the combination of 2 major criteria, 1 major and 2 minor criteria, or 3 minor criteria from the following lists. Major criteria: (1) increase in blast count; (2) evidence of cytogenetic evolution (re-appearance of a previously present or appearance of a new cytogenetic abnormality, or increase in cytogenetic burden of disease); (3) new or worsening extramedullary disease (worsening splenomegaly or extramedullary disease outside of the spleen). Minor criteria: (1) transfusion dependence; (2) significant loss of maximal response on cytopenias ≥50% decrement from maximum remission/response in granulocytes or platelets; (3) reduction in Hgb by ≥1.5g/dL from best response or from baseline as noted on complete blood count; (4) evidence of clonal evolution (molecular).
Time Frame: up to 2513 days (120 21-day treatment cycles)
Population: Full Efficacy-Evaluable Population. The confidence interval was calculated using the Brookmeyer and Crowley's method. Participants who were still alive without experiencing disease progression at the time of analysis were censored at the date of the last response assessment before the cutoff date. Participants who started a new cancer therapy before disease progression were censored at the date of last response assessment before new cancer therapy start.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemigatinib 13.5 mg
Number analyzed (Participants) | 45
months
  Investigator assessment | 73.89 [54.74 to NA] — The upper limit of the confidence interval was not estimable because too few participants had events disease progression or death.
  CRC assessment | 73.89 [29.17 to NA] — The upper limit of the confidence interval was not estimable because too few participants had events disease progression or death.

12. Secondary Outcome: Overall Survival
Description: Overall survival was defined as as the time from the first day of taking study drug until death due to any cause
Time Frame: up to 2513 days (120 21-day treatment cycles)
Population: Full Efficacy-Evaluable Population. Confidence intervals were calculated using the Brookmeyer and Crowley's method. Participants without death observed at the time of the analysis were censored at the last date known to be alive.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemigatinib 13.5 mg
Number analyzed (Participants) | 45
months | NA [54.74 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants died.

13. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related, that occurs after a participant provides informed consent. A TEAE was defined as any AE either reported for the first time or the worsening of a pre-existing event after the first dose of study drug.
Time Frame: up to 2543 days
Population: Safety Population: all enrolled participants who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Pemigatinib 13.5 mg
Number analyzed (Participants) | 47
Participants | 47

14. Secondary Outcome: Number of Participants With Any ≥Grade 3 TEAE
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related, that occurs after a participant provides informed consent. A TEAE was defined as any AE either reported for the first time or the worsening of a pre-existing event after the first dose of study drug. The severity of AEs was assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 Grades 1 through 4. Grade 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2: moderate; minimal, local, or noninvasive intervention indicated; limiting age-appropriate activities of daily living. Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living. Grade 4: life-threatening consequences; urgent intervention indicated.
Time Frame: up to 2543 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Pemigatinib 13.5 mg
Number analyzed (Participants) | 47
Participants | 39

ADVERSE EVENTS:
Time Frame: up to 2730 days
Description: Adverse events have been reported for the Safety Population, comprised of all enrolled participants who received at least 1 dose of study drug.
Arm/Group | Pemigatinib 13.5 mg
All-Cause Mortality (participants affected / at risk) | 16/47
Serious Adverse Events (participants affected / at risk) | 27/47
Other Adverse Events (participants affected / at risk) | 46/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemigatinib 13.5 mg (N=47)
Acute kidney injury (Renal and urinary disorders) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 2 (2)
Aortic stenosis (Vascular disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 2 (2)
Bladder obstruction (Renal and urinary disorders) | 1 (1)
Bladder tamponade (Renal and urinary disorders) | 1 (1)
Calciphylaxis (Metabolism and nutrition disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Corneal abscess (Infections and infestations) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1)
Erysipelas (Infections and infestations) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
General physical health deterioration (General disorders) | 1 (1)
Heart failure with preserved ejection fraction (Cardiac disorders) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (2)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Oedema genital (Reproductive system and breast disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Pneumonia aspiration (Infections and infestations) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 1 (1)
Postrenal failure (Renal and urinary disorders) | 1 (1)
Pseudomonas infection (Infections and infestations) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1)
Spinal flattening (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Stenotrophomonas infection (Infections and infestations) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Syncope (Nervous system disorders) | 2 (3)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemigatinib 13.5 mg (N=47)
Abdominal distension (Gastrointestinal disorders) | 3 (6)
Abdominal pain (Gastrointestinal disorders) | 16 (25)
Abdominal pain upper (Gastrointestinal disorders) | 7 (9)
Acute kidney injury (Renal and urinary disorders) | 3 (5)
Ageusia (Nervous system disorders) | 6 (7)
Alanine aminotransferase increased (Investigations) | 6 (11)
Alopecia (Skin and subcutaneous tissue disorders) | 26 (29)
Anaemia (Blood and lymphatic system disorders) | 16 (27)
Anxiety (Psychiatric disorders) | 5 (7)
Aphthous ulcer (Gastrointestinal disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (20)
Aspartate aminotransferase increased (Investigations) | 6 (10)
Asthenia (General disorders) | 10 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (14)
Blepharitis (Eye disorders) | 4 (4)
Blood alkaline phosphatase increased (Investigations) | 11 (14)
Blood creatinine increased (Investigations) | 8 (11)
Bronchitis (Infections and infestations) | 3 (3)
COVID-19 (Infections and infestations) | 3 (3)
Candida infection (Infections and infestations) | 3 (3)
Cataract (Eye disorders) | 5 (5)
Chills (General disorders) | 4 (5)
Confusional state (Psychiatric disorders) | 3 (3)
Conjunctival hyperaemia (Eye disorders) | 3 (3)
Conjunctivitis (Infections and infestations) | 5 (7)
Constipation (Gastrointestinal disorders) | 20 (29)
Contusion (Injury, poisoning and procedural complications) | 6 (8)
Corneal erosion (Eye disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (11)
Cystitis (Infections and infestations) | 4 (12)
Decreased appetite (Metabolism and nutrition disorders) | 16 (19)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Depression (Psychiatric disorders) | 3 (3)
Dermatitis (Skin and subcutaneous tissue disorders) | 3 (3)
Detachment of retinal pigment epithelium (Eye disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 29 (51)
Dizziness (Nervous system disorders) | 9 (16)
Dry eye (Eye disorders) | 20 (22)
Dry mouth (Gastrointestinal disorders) | 19 (20)
Dry skin (Skin and subcutaneous tissue disorders) | 12 (13)
Dysgeusia (Nervous system disorders) | 7 (7)
Dyspepsia (Gastrointestinal disorders) | 10 (11)
Dysphagia (Gastrointestinal disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (15)
Dysuria (Renal and urinary disorders) | 4 (5)
Entropion (Eye disorders) | 3 (3)
Epiretinal membrane (Eye disorders) | 3 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 16 (23)
Erysipelas (Infections and infestations) | 3 (5)
Erythema (Skin and subcutaneous tissue disorders) | 6 (7)
Eye discharge (Eye disorders) | 3 (3)
Eye pain (Eye disorders) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 4 (10)
Fatigue (General disorders) | 11 (15)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Fungal infection (Infections and infestations) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (5)
Haemorrhoids (Gastrointestinal disorders) | 5 (5)
Headache (Nervous system disorders) | 12 (15)
Hypercalcaemia (Metabolism and nutrition disorders) | 7 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (6)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 3 (4)
Hyperphosphataemia (Metabolism and nutrition disorders) | 35 (59)
Hypertension (Vascular disorders) | 5 (8)
Hypertransaminasaemia (Hepatobiliary disorders) | 4 (13)
Hyperuricaemia (Metabolism and nutrition disorders) | 3 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (6)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (5)
Hypogeusia (Nervous system disorders) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (14)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (8)
Hypophosphataemia (Metabolism and nutrition disorders) | 5 (7)
Hypotension (Vascular disorders) | 4 (6)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 3 (5)
Insomnia (Psychiatric disorders) | 5 (8)
Keratitis (Eye disorders) | 5 (6)
Lacrimation increased (Eye disorders) | 8 (9)
Leukopenia (Blood and lymphatic system disorders) | 5 (6)
Macular oedema (Eye disorders) | 3 (5)
Memory impairment (Nervous system disorders) | 6 (6)
Mouth ulceration (Gastrointestinal disorders) | 5 (6)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 (7)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (9)
Nail bed tenderness (Skin and subcutaneous tissue disorders) | 3 (4)
Nail discolouration (Skin and subcutaneous tissue disorders) | 4 (4)
Nail disorder (Skin and subcutaneous tissue disorders) | 4 (5)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 8 (8)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Nasopharyngitis (Infections and infestations) | 3 (3)
Nausea (Gastrointestinal disorders) | 17 (19)
Neck pain (Musculoskeletal and connective tissue disorders) | 5 (6)
Neuropathy peripheral (Nervous system disorders) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 4 (9)
Non-cardiac chest pain (General disorders) | 3 (3)
Oedema peripheral (General disorders) | 11 (15)
Onychalgia (Skin and subcutaneous tissue disorders) | 5 (6)
Onychoclasis (Skin and subcutaneous tissue disorders) | 4 (4)
Onycholysis (Skin and subcutaneous tissue disorders) | 8 (9)
Onychomadesis (Skin and subcutaneous tissue disorders) | 8 (8)
Oral candidiasis (Infections and infestations) | 3 (3)
Oral herpes (Infections and infestations) | 3 (3)
Oral pain (Gastrointestinal disorders) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (16)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 7 (16)
Palpitations (Cardiac disorders) | 3 (3)
Paraesthesia (Nervous system disorders) | 3 (3)
Paronychia (Infections and infestations) | 3 (3)
Pharyngitis (Infections and infestations) | 6 (6)
Photophobia (Eye disorders) | 3 (3)
Pneumonia (Infections and infestations) | 3 (4)
Pollakiuria (Renal and urinary disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (9)
Punctate keratitis (Eye disorders) | 3 (3)
Pyrexia (General disorders) | 10 (19)
Rash (Skin and subcutaneous tissue disorders) | 12 (19)
Sinusitis (Infections and infestations) | 4 (7)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 5 (5)
Skin ulcer (Skin and subcutaneous tissue disorders) | 5 (9)
Stomatitis (Gastrointestinal disorders) | 21 (51)
Subretinal fluid (Eye disorders) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (8)
Tremor (Nervous system disorders) | 3 (3)
Trichiasis (Eye disorders) | 7 (8)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Urinary tract infection (Infections and infestations) | 7 (11)
Vision blurred (Eye disorders) | 10 (10)
Visual acuity reduced (Eye disorders) | 3 (3)
Vitamin D deficiency (Metabolism and nutrition disorders) | 5 (6)
Vomiting (Gastrointestinal disorders) | 7 (19)
Weight decreased (Investigations) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2023-07-13): https://cdn.clinicaltrials.gov/large-docs/72/NCT03011372/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-24): https://cdn.clinicaltrials.gov/large-docs/72/NCT03011372/SAP_001.pdf